CLINICAL TRIAL: NCT04290234
Title: The Influence of Childhood Maltreatment on Cognitive and Reactive Fear
Brief Title: Childhood Trauma and Escape Decision Dynamics
Acronym: TEDDY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Prof. Dean Mobbs (Unknown)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor for Psychiatry, University of Oldenburg
Other Study IDs: TEDDY
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Child Abuse; Fear
Keywords: cognitive fear; fMRI; reactive fear

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-medicated healthy adults with childhood maltreatment: The 25-item retrospective Childhood Trauma Questionnaire (CTQ) will be administered to assess history of abuse and neglect. The CTQ measures five types of maltreatment: emotional, physical, and sexual abuse and emotional and physical neglect.
  Interventions: Other: fMRI assessment of cognitive and reactive fear

INTERVENTIONS:
Other: fMRI assessment of cognitive and reactive fear — An fMRI paradigm will be used to probe how childhood maltreatment may modulate the defensive survival circuitry that facilitates escape decisions when subjects encounter fast- or slow-attacking threats.

SUMMARY:
The purpose of this study is to evaluate the effects of childhood maltreatment on cognitive and reactive fear.

DETAILED DESCRIPTION:
Childhood maltreatment dramatically increases the risk for psychiatric disorders accompanied by profound difficulties in social interactions. However, it is still unclear how childhood maltreatment affects social interactions in adulthood. In this study, we examine how childhood maltreatment may modulate threat sensitivity assessed by the distance at which an individual flees from an approaching threat. While rapid escape decisions rely on "reactive fear" circuits, slower escape decisions are associated with "cognitive fear" circuits. Based on previous observations of altered early sensory processing, we expect that childhood maltreatment affects both cognitive and reactive fear circuits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with varying levels of childhood maltreatment

Exclusion Criteria:

* current psychiatric illness
* current psychiatric medication or psychotherapy
* MRI contraindication (e.g. metal in body, claustrophobia)
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a community sample and childhood maltreatment will be assessed with the Childhood Trauma Questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-11-17 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Neural responses in the flight initiation distance (FID) task | fMRI paradigm with an average duration of 45 minutes
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal in a flight initiation distance (FID) task, involving fast-, medium- and slow-attacking virtual predators that elicit distinct activations in the reactive and cognitive fear circuits. Blood-oxygen-level-dependent signals to different predator velocities will be analyzed. Analyses will focus on regions-of-interest associated with the processing of cognitive fear (ventromedial prefrontal cortex, posterior cingulate cortex, hippocampus, and basolateral amygdala) and reactive fear (midbrain periaqueductal gray, central amygdala, hypothalamus, and the midcingulate cortex). To examine effects of childhood maltreatment, regression analyses with Childhood Trauma Questionnaire scores will be conducted on the second level.
Flight distance in the flight initiation distance (FID) task | fMRI paradigm with an average duration of 45 minutes
  Associations between the flight distance in the FID task and childhood maltreatment will be analyzed using regression analyses with Childhood Trauma Questionnaire scores. Behavioral data will be correlated with fMRI data of the FID task.
Difficulty ratings in the flight initiation distance (FID) task | fMRI paradigm with an average duration of 45 minutes
  Associations between the difficulty ratings in the FID task and childhood maltreatment will be analyzed using regression analyses with Childhood Trauma Questionnaire scores. Behavioral data will be correlated with fMRI data of the FID task.
Confidence ratings in the flight initiation distance (FID) task | fMRI paradigm with an average duration of 45 minutes
  Associations between the confidence ratings in the FID task and childhood maltreatment will be analyzed using regression analyses with Childhood Trauma Questionnaire scores. Behavioral data will be correlated with fMRI data of the FID task.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Scheele, PhD, Principal Investigator — University of Bonn
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided